CLINICAL TRIAL: NCT02377349
Title: Immunogenicity and Safety Study of GSK Biologicals' dTpa Vaccine, Boostrix™ (263855) in Pregnant Women
Brief Title: Immunogenicity and Safety Study of GlaxoSmithKline (GSK) Biologicals' Boostrix™ Vaccine in Pregnant Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 116945; 2014-001119-38 (EudraCT Number)
Record Dates: First submitted 2015-02-26; First posted 2015-03-03 (Estimated); Results first posted 2019-01-28 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Diphtheria-Tetanus-acellular Pertussis Vaccines
MeSH Terms: interventions — Boostrix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dTpa Group (Experimental): This group will consist of pregnant women who will receive a single dose of Boostrix™ at 27-36 weeks (i.e. completed 27 weeks until 36 weeks) of gestation (Visit 1) and will receive a dose of the placebo post-delivery (within 72 hours).
  Interventions: Biological: Boostrix™; Drug: Saline placebo
- Control Group (Placebo Comparator): This group will consist of pregnant women who will receive a single dose of placebo at 27-36 weeks (i.e. completed 27 weeks until 36 weeks) of gestation (Visit 1) and will receive a dose of Boostrix™ post-delivery (within 72 hours).
  Interventions: Biological: Boostrix™; Drug: Saline placebo

INTERVENTIONS:
Biological: Boostrix™ — One dose administered intramuscularly in the deltoid muscle of the non-dominant arm.
Drug: Saline placebo — One dose administered intramuscularly in the deltoid muscle of the non-dominant arm.

SUMMARY:
The purpose of this study is to assess the immunogenicity and safety of Boostrix™ when compared to a placebo given during 27-36 weeks of gestation in healthy women aged 18-45 years. Infants born to mothers enrolled in this study will be followed-up in two separate clinical studies: 201330 [DTPA (BOOSTRIX)-048 PRI] and 201334 [DTPA (BOOSTRIX)-049 BST: 048].

DETAILED DESCRIPTION:
The protocol was amended to include Spain in the study. The reasons for the Spain-specific amendment are listed below:

* Based on the feedback from the Spanish Ethics Committee, the evaluation related to the acceptance of cocooning was added in the protocol.
* The objectives and endpoints to include cocooning were added in the protocol.
* The eligibility criteria for participation of household contacts were defined in the protocol.
* The study procedures for household contacts were included.

ELIGIBILITY:
Inclusion Criteria for study subjects:

* Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Written informed consent obtained from the subject prior to performing any study specific procedure, as per local regulations.
* A healthy pregnant woman between, and including, 18 and 45 years of age at the time of screening.
* Pregnant subjects at 27 0/7-36 6/7 weeks (completed 27 weeks but not 37 weeks) of gestation at the time of vaccination (Visit 1), as established by ultrasound examination.
* Not at high risk for complications, as determined by the obstetrical algorithm for identification of eligible subjects and the Obstetrical Risk Assessment Form.
* No significant foetal abnormalities, as observed by the level II ultrasound testing conducted after 18 weeks of gestation.
* Nuchal translucency scan, serum testing and any other prenatal tests, if conducted, should suggest normal pregnancy.
* Willing to have the infant born immunised with Infanrix hexa and Prevenar 13, as per national recommendations, in the follow-up clinical studies DTPA (BOOSTRIX)-048 PRI and DTPA (BOOSTRIX)-049 BST: 048.
* Subjects who do not plan to give their child for adoption or place the child in care.

Inclusion criteria for household contacts in Spain:

* Household contacts living in the same house as that of the infant.
* Household contacts or parent(s)/LAR(s) of the household contacts who, in the opinion of the investigator, can and will comply with the requirements of the protocol (e.g. reporting of SAEs).
* Written informed consent obtained from the household contacts or the parent(s)/LAR(s) prior to vaccination, as per local regulations.
* Household contacts who are eligible to receive a booster dose of DTP-containing vaccine according to the Summary of Product Characteristics (SmPC) of Boostrix and according to the local governmental recommendations in Spain.
* Female household contacts of non-childbearing potential may be enrolled in the study.

  - Non-childbearing potential is defined as pre-menarche, current tubal ligation, hysterectomy, ovariectomy or post-menopause.
* Female household contacts of childbearing potential may be enrolled in the study , if the household contact

  * has practiced adequate contraception for 30 days prior to vaccination,
  * has a negative pregnancy test on the day of vaccination and
  * has agreed to continue adequate contraception for 2 months after receiving the vaccine dose.

Exclusion Criteria for study subjects:

* Subjects diagnosed with multiple pregnancies (twins, triplets etc.).
* Previous vaccination containing diphtheria, tetanus or pertussis antigens or diphtheria and tetanus toxoids at any time during the current pregnancy.
* Women with co-morbid medical or obstetric conditions that in the opinion of the investigator have the potential to complicate the pregnancy course and outcomes.
* Gestational diabetes as determined by glucose tolerance test conducted after 20 weeks of gestation, as per local recommendations of the country.
* History of early onset (<34 weeks of gestation) of eclampsia/pre-eclampsia in previous pregnancy.
* History of major congenital anomalies in previous pregnancies.
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine anytime during the current pregnancy or planned use during the study period.
* Any medical condition that in the judgment of the investigator would make intramuscular injection unsafe.
* Chronic administration of immunosuppressants or other immune-modifying drugs during the period starting six months prior to the first vaccine. For corticosteroids, this will mean prednisone ≥20 mg/day, or equivalent. Inhaled and topical steroids are allowed.
* Administration of long-acting immune-modifying drugs at any time during the study period.
* Planned administration/administration of a vaccine not foreseen by the study protocol in the period within the period starting 30 days before and 30 days after the dose of vaccine with the exception of seasonal influenza vaccine that can be administered anytime during the study period.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product (pharmaceutical product or device).
* Serious underlying medical condition [e.g., immunosuppressive disease or therapy, human immunodeficiency virus infection, collagen vascular disease, epilepsy, diabetes mellitus, chronic hypertension, moderate to severe asthma, lung/heart disease, liver/kidney disease, infections including TORCHES (toxoplasmosis, rubella, cytomegalovirus, herpes simplex, syphilis) infections].
* History of an encephalopathy of unknown aetiology, occurring within 7 days following previous vaccination with pertussis-containing vaccine.
* History of transient thrombocytopenia or neurological complications (for convulsions or hypotonic-hyporesponsive episodes) following an earlier immunisation against diphtheria and/or tetanus
* Significant mental illness (e.g. schizophrenia, psychosis and major depression).
* Family history (first degree relatives only) of congenital anomalies, recurrent pregnancy losses (two or more consecutive losses) and unexplained neonatal death(s) in the subject.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine.
* History of febrile illness within the past 72 hours.
* History of physician-diagnosed or laboratory-confirmed pertussis within the past five years.
* Anything that would prevent subject from completing the study or put the subject at risk, as determined by the investigator.
* Acute disease and/or fever at the time of enrolment.

  * Fever is defined as temperature ≥ 37.5°C /99.5°F for oral, axillary or tympanic route, or ≥ 38.0°C /100.4°F on rectal route.
  * Subjects with a minor illness (such as mild diarrhoea, mild upper respiratory infection) without fever may be enrolled at the discretion of the investigator.
* Administration of immunoglobulins and/or any blood products within the 3 months preceding the dose of study vaccine, or planned administration during the study period, with the exception of anti-D (Rh)-immunoglobulin.
* History of chronic excessive alcohol consumption and/or drug abuse.

Exclusion criteria for household contacts in Spain:

* Child in care.
* Concurrently participating in another clinical study, at any time during the study period, in which the household contact has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine within 30 days preceding the dose of study vaccine, or planned use during the study period.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine.
* History of an encephalopathy of unknown aetiology, occurring within 7 days following previous vaccination with pertussis-containing vaccine.
* Acute disease and/or fever at the time of enrolment.

  * Fever is defined as temperature ≥ 37.5°C /99.5°F for oral, axillary or tympanic route, or ≥ 38.0°C /100.4°F on rectal route. The preferred route of recording temperature will be axillary in household contacts.
  * Household contacts with a minor illness (such as mild diarrhoea, mild upper respiratory infection) without fever may be enrolled at the discretion of the investigator.
* Anything that would put the household contact at risk, as determined by the investigator.
* Pregnant or lactating household contacts.
* Household contacts planning to become pregnant or planning to discontinue contraceptive precautions prior to 2 months post-vaccination.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 688 (Actual)
Dates: Start 2015-10-14 (Actual); Primary Completion 2017-08-14 (Actual); Study Completion 2017-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (30):
- Australia (3):
  - GSK Investigational Site, Carlton, Victoria
  - GSK Investigational Site, Fitzroy, Victoria
  - GSK Investigational Site, Parkville, Victoria
- Canada (5):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Greater Sudbury, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Mount Royal, Quebec
- Czechia (4):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Hradec Králové
  - GSK Investigational Site, Ostrava - Vitkovice
  - GSK Investigational Site, Prague
- Finland (5):
  - GSK Investigational Site, Kokkola
  - GSK Investigational Site, Oulu
  - GSK Investigational Site, Seinäjoki
  - GSK Investigational Site, Tampere
  - GSK Investigational Site, Turku
- Italy (3):
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Novara, Piedmont
  - GSK Investigational Site, Turin, Piedmont
- Spain (10):
  - GSK Investigational Site, Málaga, Andalusia
  - GSK Investigational Site, Antequera/Málaga
  - GSK Investigational Site, Aravaca
  - GSK Investigational Site, Boadilla del Monte
  - GSK Investigational Site, Burgos
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Majadahonda (Madrid)
  - GSK Investigational Site, Móstoles
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Seville

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Background] Perrett KP, Halperin SA, Nolan T, Martinez Pancorbo C, Tapiero B, Martinon-Torres F, Stranak Z, Virta M, Vanderkooi OG, Kosina P, Encinas Pardilla MB, Cristobal Garcia I, Zuccotti GV, Kostanyan L, Meyer N, Ceregido MA, Cheuvart B, Kuriyakose SO, Marcos Fernandez M, Rodriguez Zambrano MA, Martin Garcia A, Asenjo de la Fuente JE, Camacho Marin MD, de la Calle Fernandez-Miranda M, Romero Espinar Y, Marchisio PG, Manzoni P, Mesaros N. Immunogenicity, transplacental transfer of pertussis antibodies and safety following pertussis immunization during pregnancy: Evidence from a randomized, placebo-controlled trial. Vaccine. 2020 Feb 18;38(8):2095-2104. doi: 10.1016/j.vaccine.2019.10.105. Epub 2019 Nov 24. PMID 31776029

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 725 pregnant subjects were screened of which 690 were randomized to 2 groups. Of these, 2 subjects were withdrawn before vaccination. Therefore 688 subjects were enrolled: 1 subject was excluded from the statistical analysis, leaving 687 subjects that comprised the Total Vaccinated cohort.
Pre-assignment Details: Safety was assessed for infants born to vaccinated subjects as well as safety of dTap vaccination in the vaccinated pregnant subjects. There was also an assessment of the acceptance rate of a single dose of Boostrix among 723 eligible household contacts of the infants born to pregnant women enrolled in Spain, as part of an assessment of cocooning.
Groups:
- dTpa Group - Mother: This group consisted of pregnant women who received a single dose of Boostrix at 27-36 weeks (i.e. 27 weeks until 36 completed weeks) of gestation (Visit 1) and received a dose of the placebo post-delivery (within 72 hours).
- Control Group - Mother: This group consisted of pregnant women who received a single dose of placebo at 27-36 weeks (i.e. 27 weeks until 36 completed weeks) of gestation (Visit 1) and received a dose of Boostrix post-delivery (within 72 hours).
Period: Overall Study
Arm/Group | dTpa Group - Mother | Control Group - Mother
Started | 341 | 346
Completed | 325 | 335
Not Completed | 16 | 11
Not completed — Serious Adverse Event | 1 | 0
Not completed — Protocol Violation | 3 | 2
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Lost to follow-up (partial vaccination) | 1 | 0
Not completed — Lost to follow-up (complete vaccination) | 6 | 5
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | dTpa Group - Mother | Control Group - Mother | Total
Number analyzed (Participants) | 341 | 346 | 687
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.7 (4.4) | 32.5 (4.3) | 32.6 (4.35)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 341 | 346 | 687
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African Heritage / African American | 3 | 9 | 12
  American Indian or Alaskan Native | 2 | 0 | 2
  Asian - Central/South Asian Heritage | 3 | 0 | 3
  Asian - East Asian Heritage | 4 | 1 | 5
  Asian - Japanese Heritage | 1 | 0 | 1
  Asian - South East Asian Heritage | 1 | 1 | 2
  White - Arabic / North African Heritage | 3 | 7 | 10
  White - Caucasian / European Heritage | 314 | 319 | 633
  Unspecified | 10 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: Antibody Concentrations Against Pertussis Toxoid Antigen (Anti-PT), Filamentous Haemagglutinin Antigen (Anti-FHA) and Pertactin Antigen (Anti-PRN) in Cord Blood Samples
Description: Antibody concentrations were assessed by Enzyme-linked immunosorbent assay (ELISA), tabulated as Geometric Mean Concentrations (GMCs) and expressed in International units per mililiter (IU/mL) for the following assay cut-offs: 2.693 IU/mL for anti-PT, 2.046 IU/mL for anti-FHA and 2.187 IU/mL for anti-PRN.
Time Frame: At delivery - Visit 3 (anytime after 28 weeks of gestation)
Population: The analysis was done on the According to protocol cohort for immunogenicity , which included all evaluable subjects who complied with the vaccine administration, who had cord blood collected at least 21 days post-vaccination and for whom data concerning antibodies against at least 1 study vaccine antigen component at Visit 3 were available.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | dTpa Group - Mother | Control Group - Mother
Number analyzed (Participants) | 291 | 292
IU/mL
  Anti-PT: number analyzed (Participants) | 290 | 292
  Anti-PT | 46.9 [41.2 to 53.3] | 5.5 [4.8 to 6.3]
  Anti-FHA | 366.1 [329 to 407.3] | 22.7 [19.7 to 26.2]
  Anti-PRN: number analyzed (Participants) | 290 | 291
  Anti-PRN | 301.8 [250.9 to 362.9] | 14.6 [12.1 to 17.7]
Statistical Analysis 1: Comparison: dTpa Group - Mother vs Control Group - Mother; GMC ratio between groups (dTpa Group-Mother/Control Group-Mother) to demonstrate that maternally transferred antibodies against pertussis in the dTpa Group-Mother was superior to that in the Control Group-mother, in the cord blood sample at the time of delivery; Test type: Superiority — Criterion: The lower limit (LL) of the 95% confidence interval (CI) of the GMC ratio [dTpa Group-Mother/Control Group-Mother] for anti-PT antibodies was greater than or equal to (≥) 1.5; 2-sample t-test; The CI of the group GMC ratio were computed using two-sample t-test assuming heterogeneity of variance; GMC ratio = 8.47, 95% CI 2-sided [7.02 to 10.2]
Statistical Analysis 2: Comparison: dTpa Group - Mother vs Control Group - Mother; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — Criterion: The lower limit (LL) of the 95% confidence interval (CI) of the GMC ratio [dTpa Group-Mother/Control Group-Mother] for anti-FHA antibodies was greater than or equal to (≥) 1.5; 2-sample t-test; The CI of the group GMC ratio were computed using two-sample t-test assuming heterogeneity of variance; GMC ratio = 16.11, 95% CI 2-sided [13.48 to 19.24]
Statistical Analysis 3: Comparison: dTpa Group - Mother vs Control Group - Mother; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — Criterion: The lower limit (LL) of the 95% confidence interval (CI) of the GMC ratio [dTpa Group-Mother/Control Group-Mother] for anti-PRN antibodies was greater than or equal to (≥) 1.5; 2-sample t-test; The CI of the group GMC ratio were computed using two-sample t-test assuming heterogeneity of variance; GMC ratio = 20.65, 95% CI 2-sided [15.86 to 26.88]

2. Secondary Outcome: Percentage of Subjects by Pregnancy Outcomes
Description: Pregnancy outcomes included live birth with no congenital anomalies, live birth with congenital anomalies, still birth with no congenital anomalies, still birth with congenital anomalies, elective termination with no congenital anomalies and elective termination with congenital anomalies. No subjects with still birth or elective termination of infant were reported.
Time Frame: From Day 0 (Visit 1) to Month 2 (Visit 4, end of the study).
Population: This analysis was performed on the Total Vaccinated cohort (TVC) which included all subjects with the study vaccine administration documented.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | dTpa Group - Mother | Control Group - Mother
Number analyzed (Participants) | 341 | 346
Percentage of subjects
  Live infant No apparent congenital anomaly | 97.4 [95 to 98.8] | 97.4 [95.1 to 98.8]
  Live infant congenital anomaly | 2.6 [1.2 to 5] | 2.3 [1 to 4.5]
  Lost to follow-up | 0 [0 to 1.1] | 0.3 [0 to 1.6]

3. Secondary Outcome: Percentage of Subjects With Listed Pregnancy/Neonate Related Adverse Events of Interest
Description: Listed pregnancy-related adverse events of interest/ neonate-related events of interest included gestational diabetes, pregnancy-related hypertension, premature rupture of mem-branes, preterm premature rupture of membranes, premature labour, premature uterine contractions, intrauterine growth restriction/poor foetal growth, pre-eclampsia, eclampsia, vaginal or intrauterine haemorrhage, maternal death, preterm birth, neonatal death, small for gestational age, neonatal hypoxic ischaemic encephalopathy and failure to thrive/growth deficiency were reported.
Time Frame: From Day 0 (Visit 1) to Month 2 post-delivery (Visit 4, end of the study).
Population: This analysis was performed on the TVC which included all subjects with the study vaccine administration documented.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | dTpa Group - Mother | Control Group - Mother
Number analyzed (Participants) | 341 | 346
Percentage of subjects
  Intrauterine growth restriction/poor foetal growth | 1.5 [0.5 to 3.4] | 0.6 [0.1 to 2.1]
  Pre-eclampsia | 0.3 [0 to 1.6] | 1.4 [0.5 to 3.3]
  Pregnancy-related hypertension | 1.2 [0.3 to 3] | 1.4 [0.5 to 3.3]
  Premature labour | 3.8 [2 to 6.4] | 3.2 [1.6 to 5.6]
  Premature rupture of membranes | 3.8 [2 to 6.4] | 4.3 [2.4 to 7]
  Premature uterine contractions | 0.6 [0.1 to 2.1] | 0.9 [0.2 to 2.5]
  Preterm birth | 3.2 [1.6 to 5.7] | 2.6 [1.2 to 4.9]
  Preterm premature rupture of membranes | 1.2 [0.3 to 3] | 2 [0.8 to 4.1]
  Small for gestational age | 0.6 [0.1 to 2.1] | 0.6 [0.1 to 2.1]
  Vaginal or intrauterine haemorrhage | 2.6 [1.2 to 5] | 2.9 [1.4 to 5.3]

4. Secondary Outcome: Percentage of Seroprotected Subjects Against Diphteria Antigen (Anti-D), Tetanus Antigen (Anti-T) and of Seropositive Subjects Against Anti-PT, Anti-FHA and Anti-PRN
Description: A seroprotected subject against diphteria and tetanus was a subject with antibody concentration ≥ 0.1 IU/mL. A seropositive subject was a subjects with antibody concentration ≥ 2.693 IU/mL for anti-PT, ≥ 2.046 IU/mL for anti-FHA and ≥ 2.187 IU/mL for anti-PRN.
Time Frame: One month post vaccination (Day 30) during pregnancy
Population: The analysis was done on the According to protocol cohort for immunogenicity , which included all evaluable subjects who complied with the vaccine administration and for whom data concerning antibodies against at least 1 study vaccine antigen component at Visit 2 were available.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | dTpa Group - Mother | Control Group - Mother
Number analyzed (Participants) | 290 | 292
Percentage of subjects
  Anti-D: number analyzed (Participants) | 290 | 289
  Anti-D | 97.6 [95.1 to 99] | 70.6 [65 to 75.8]
  Anti-T | 100 [98.7 to 100] | 96.6 [93.8 to 98.3]
  Anti-PT: number analyzed (Participants) | 289 | 292
  Anti-PT | 98.6 [96.5 to 99.6] | 61.3 [55.5 to 66.9]
  Anti-FHA: number analyzed (Participants) | 290 | 291
  Anti-FHA | 100 [98.7 to 100] | 94.5 [91.2 to 96.8]
  Anti-PRN: number analyzed (Participants) | 290 | 291
  Anti-PRN | 100 [98.7 to 100] | 84.5 [79.9 to 88.5]

5. Secondary Outcome: Anti-D, Anti-T, Anti-PT, Anti-FHA and Anti-PRN Antibody Concentrations
Description: Antibody concentrations were determined by ELISA, tabulated as GMCs and expressed in IU/mL.
Time Frame: One month post vaccination (Day 30) during pregnancy
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | dTpa Group - Mother | Control Group - Mother
Number analyzed (Participants) | 290 | 292
IU/mL
  Anti-D: number analyzed (Participants) | 290 | 289
  Anti-D | 2.19 [1.87 to 2.57] | 0.23 [0.19 to 0.27]
  Anti-T | 8.43 [7.72 to 9.2] | 0.98 [0.86 to 1.11]
  Anti-PT: number analyzed (Participants) | 289 | 292
  Anti-PT | 45.6 [40.4 to 51.5] | 4.1 [3.6 to 4.6]
  Anti-FHA: number analyzed (Participants) | 290 | 291
  Anti-FHA | 317.5 [285 to 353.8] | 15 [13.1 to 17.2]
  Anti-PRN: number analyzed (Participants) | 290 | 291
  Anti-PRN | 283.6 [237.1 to 339.1] | 10.5 [8.7 to 12.5]

6. Secondary Outcome: Percentage of Subjects With Vaccine Response to Anti-D and Anti-T
Description: Vaccine response for anti-D and anti-T was defined as:
  for initially seronegative subjects (S-) with pre-vaccination concentration below cut-off: < 0.1 IU/mL) was an antibody concentration at least four times the assay cut-off (post-vaccination concentration ≥ 0.4 IU/mL); for initially seropositive subjects (S+) with pre-vaccination concentration ≥ 0.1 IU/mL): an increase in antibody concentrations of at least four times the pre-vaccination concentration.
Time Frame: One month post vaccination (Day 30) during pregnancy
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | dTpa Group - Mother | Control Group - Mother
Number analyzed (Participants) | 288 | 291
Percentage of subjects
  Anti-D, S-: number analyzed (Participants) | 103 | 83
  Anti-D, S- | 64.1 [54 to 73.3] | 0 [0 to 4.3]
  Anti-D, S+: number analyzed (Participants) | 184 | 205
  Anti-D, S+ | 75 [68.1 to 81.1] | 0 [0 to 1.8]
  Anti-D, Total: number analyzed (Participants) | 287 | 288
  Anti-D, Total | 71.1 [65.5 to 76.3] | 0 [0 to 1.3]
  Anti-T, S-: number analyzed (Participants) | 12 | 10
  Anti-T, S- | 100 [73.5 to 100] | 0 [0 to 30.8]
  Anti-T, S+: number analyzed (Participants) | 276 | 281
  Anti-T, S+ | 67.8 [61.9 to 73.2] | 0 [0 to 1.3]
  Anti-T, Total | 69.1 [63.4 to 74.4] | 0 [0 to 1.3]

7. Secondary Outcome: Percentage of Subjects With Vaccine Response to Anti-PT, Anti-FHA and Anti-PRN
Description: Vaccine response to PT, FHA and PRN antigens is defined as: for subjects with pre-vaccination antibody concentration below the assay cut-off (S-), post-vaccination anti-body concentration ≥ 4 times the assay cut-off; for subjects with pre-vaccination antibody concentration between the assay cut-off and below 4 times the assay cut-off (S+), post-vaccination antibody concentration ≥ 4 times the pre-vaccination antibody concentration, and for subjects with pre-vaccination antibody concentration ≥4 times the assay cut-off (S+), post-vaccination antibody concentration ≥2 times the pre-vaccination antibody concentration.
Time Frame: One month post vaccination (Day 30) during pregnancy
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | dTpa Group - Mother | Control Group - Mother
Number analyzed (Participants) | 288 | 291
Percentage of subjects
  Anti-PT, S-: number analyzed (Participants) | 121 | 107
  Anti-PT, S- | 82.6 [74.7 to 88.9] | 0.9 [0 to 5.1]
  Anti-PT, S+ (<4 cut-off): number analyzed (Participants) | 108 | 117
  Anti-PT, S+ (<4 cut-off) | 90.7 [83.6 to 95.5] | 0 [0 to 3.1]
  Anti-PT, S+ (≥4 cut-off): number analyzed (Participants) | 58 | 67
  Anti-PT, S+ (≥4 cut-off) | 93.1 [83.3 to 98.1] | 3 [0.4 to 10.4]
  Anti-PT, Total: number analyzed (Participants) | 287 | 291
  Anti-PT, Total | 87.8 [83.4 to 91.4] | 1 [0.2 to 3]
  Anti-FHA, S-: number analyzed (Participants) | 16 | 16
  Anti-FHA, S- | 100 [79.4 to 100] | 0 [0 to 20.6]
  Anti-FHA, S+ (<4 cut-off): number analyzed (Participants) | 84 | 65
  Anti-FHA, S+ (<4 cut-off) | 100 [95.7 to 100] | 0 [0 to 5.5]
  Anti-FHA, S+ (≥4 cut-off): number analyzed (Participants) | 188 | 209
  Anti-FHA, S+ (≥4 cut-off) | 89.9 [84.7 to 93.8] | 1.9 [0.5 to 4.8]
  Anti-FHA, Total: number analyzed (Participants) | 288 | 290
  Anti-FHA, Total | 93.4 [89.9 to 96] | 1.4 [0.4 to 3.5]
  Anti-PRN, S-: number analyzed (Participants) | 45 | 43
  Anti-PRN, S- | 86.7 [73.2 to 94.9] | 0 [0 to 8.2]
  Anti-PRN, S+ (<4 cut-off): number analyzed (Participants) | 98 | 86
  Anti-PRN, S+ (<4 cut-off) | 95.9 [89.9 to 98.9] | 0 [0 to 4.2]
  Anti-PRN, S+ (≥4 cut-off): number analyzed (Participants) | 145 | 161
  Anti-PRN, S+ (≥4 cut-off) | 86.2 [79.5 to 91.4] | 1.2 [0.2 to 4.4]
  Anti-PRN Total: number analyzed (Participants) | 288 | 290
  Anti-PRN Total | 89.6 [85.5 to 92.9] | 0.7 [0.1 to 2.5]

8. Secondary Outcome: Percentage of Seropositive Subjects Against Anti-PT, Anti-FHA and Anti-PRN in the Cord Blood Samples
Description: For this assay the anti-PT, anti-FHA and anti-PRN seropositivity status was determined from the cord blood samples. The seropositivity cut-offs were the following: 2.693 IU/mL for anti-PT, 2.046 IU/mL for anti-FHA and 2.187 IU/mL for anti-PRN.
Time Frame: At delivery - Visit 3 (anytime after 27 eligible weeks of gestation)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | dTpa Group - Mother | Control Group - Mother
Number analyzed (Participants) | 291 | 292
Percentage of subjects
  Anti-PT: number analyzed (Participants) | 290 | 292
  Anti-PT | 98.6 [96.5 to 99.6] | 68.8 [63.2 to 74.1]
  Anti-FHA | 100 [98.7 to 100] | 96.6 [93.8 to 98.3]
  Anti-PRN: number analyzed (Participants) | 290 | 291
  Anti-PRN | 99.7 [98.1 to 100] | 88 [83.7 to 91.5]

9. Secondary Outcome: Percentage of Subjects With Solicited Local Adverse Events (AEs)
Description: Assessed solicited local symptoms were pain, redness and swelling. "Any" = any report of the specified symptom irrespective of intensity grade. Dose 1 = pregnancy dose at Day 0 - Visit 1, Dose 2 = post-delivery dose at birth - Visit 3.
Time Frame: During the 8-day (Day 0-Day 7) follow-up period after vaccination during pregnancy
Population: The analysis was done on the TVC, which included all subjects with the study vaccine administration documented and who had returned their diary cards.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | dTpa Group - Mother | Control Group - Mother
Number analyzed (Participants) | 335 | 343
Percentage of subjects
  Any Pain, Dose 1 | 86.3 [82.1 to 89.8] | 14.6 [11 to 18.8]
  Any Redness (mm), Dose 1 | 28.7 [23.9 to 33.8] | 12.8 [9.5 to 16.8]
  Any Swelling (mm), Dose 1 | 25.1 [20.5 to 30.1] | 3.5 [1.8 to 6]
  Any Pain, Dose 2: number analyzed (Participants) | 324 | 330
  Any Pain, Dose 2 | 12.7 [9.2 to 16.8] | 62.7 [57.3 to 68]
  Any Redness (mm), Dose 2: number analyzed (Participants) | 324 | 330
  Any Redness (mm), Dose 2 | 10.5 [7.4 to 14.4] | 29.7 [24.8 to 34.9]
  Any Swelling (mm), Dose 2: number analyzed (Participants) | 324 | 330
  Any Swelling (mm), Dose 2 | 5.2 [3.1 to 8.3] | 26.4 [21.7 to 31.5]

10. Secondary Outcome: Percentage of Subjects With Solicited General AEs
Description: Assessed solicited general symptoms were fatigue, gastrointestinal symptoms (nausea, vomiting, diarrhoea and/or abdominal pain), headache and fever [defined as oral, axillary or tympanic temperature ≥ 37.5 degrees Celsius (°C) or rectal temperature ≥ 38.0 °C]. "Any" = any report of the specified symptom irrespective of intensity grade. Dose 1 = pregnancy dose at Day 0 - Visit 1, Dose 2 = post-delivery dose at birth - Visit 3.
Time Frame: During the 8-day (Day 0-Day 7) follow-up period after vaccination during pregnancy
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | dTpa Group - Mother | Control Group - Mother
Number analyzed (Participants) | 335 | 342
Percentage of subjects
  Any Fatigue, Dose 1 | 43.6 [38.2 to 49.1] | 36.3 [31.2 to 41.6]
  Any Gastrointestinal symptom, Dose 1 | 17.9 [14 to 22.4] | 15.2 [11.6 to 19.5]
  Any Headache, Dose 1 | 24.8 [20.2 to 29.8] | 22.8 [18.5 to 27.6]
  Any Temperature/(Axillary) (°C), Dose 1 | 1.2 [0.3 to 3] | 0.9 [0.2 to 2.5]
  Any Fatigue, Dose 2: number analyzed (Participants) | 324 | 331
  Any Fatigue, Dose 2 | 40.1 [34.7 to 45.7] | 46.2 [40.8 to 51.8]
  Any Gastrointestinal symptom, Dose 2: number analyzed (Participants) | 324 | 331
  Any Gastrointestinal symptom, Dose 2 | 9.9 [6.9 to 13.7] | 12.7 [9.3 to 16.8]
  Any Headache, Dose 2: number analyzed (Participants) | 324 | 331
  Any Headache, Dose 2 | 23.1 [18.7 to 28.1] | 23.6 [19.1 to 28.5]
  Any Temperature/(Axillary) (°C), Dose 2: number analyzed (Participants) | 324 | 331
  Any Temperature/(Axillary) (°C), Dose 2 | 4.6 [2.6 to 7.5] | 9.1 [6.2 to 12.7]

11. Secondary Outcome: Percentage of Subjects With Unsolicited AEs
Description: An unsolicited AE was any AE that was not solicited using a subject diary and that was spontaneously communicated by the subject. Also any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms was reported as an unsolicited adverse event. Dose 1 = pregnancy dose at Day 0 - Visit 1, Dose 2 = post-delivery dose at birth - Visit 3.
Time Frame: Within 31 days (Day 0 - Day 30) after each vaccination
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | dTpa Group - Mother | Control Group - Mother
Number analyzed (Participants) | 341 | 346
Percentage of subjects
  Any unsolicited AE, Dose 1 | 38.7 [33.5 to 44.1] | 35.5 [30.5 to 40.8]
  Any unsolicited AE, Dose 2: number analyzed (Participants) | 336 | 342
  Any unsolicited AE, Dose 2 | 30.7 [25.8 to 35.9] | 32.2 [27.2 to 37.4]

12. Secondary Outcome: Percentage of Infants With Unsolicited AEs
Description: An unsolicited AE was any AE that was not solicited using a subject diary and that was spontaneously communicated by the subject. Also any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms was reported as an unsolicited adverse event.
Time Frame: From delivery to Month 2 post delivery (Visit 4, end of the study).
Population: The analysis was done on the TVC of Mother, which included all subjects with the study vaccine administration documented and who had returned their diary cards.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Groups:
- dTpa Group - Infant: This group consisted of infants born to mothers (from dTpa Group Mother) who received a dose of Boostrix during pregnancy.
- Control Group - Infnat: This group consisted of infants born to mothers (from Control Group Mother) who received a dose of placebo during pregnancy.
Arm/Group | dTpa Group - Infant | Control Group - Infnat
Number analyzed (Participants) | 341 | 346
Percentage of subjects | 26.4 [21.8 to 31.4] | 22.3 [18.0 to 27.0]

13. Secondary Outcome: Number of Subjects With Serious AEs (SAEs)
Description: A SAE was any untoward medical occurrence that resulted in death, was life threatening, required hospitalization or prolongation of hospitalization, resulted in disability/incapacity or a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: From Day 0 (Visit 1) to Month 2 (Visit 4, end of the study).
Population: The analysis was done on the TVC, which included all subjects with the study vaccine administration documented.
Measure: Count of Participants; unit: Participants
Groups:
- Control Group - Infant: This group consisted of infants born to mothers (from Control Group Mother) who received a dose of placebo during pregnancy
- Household Group: This group consisted of eligible household contacts of the infants born to pregnant women enrolled in Spain who received a single dose of Boostrix anytime during the study.
Arm/Group | dTpa Group - Mother | Control Group - Mother | dTpa Group - Infant | Control Group - Infant | Household Group
Number analyzed (Participants) | 341 | 346 | 341 | 346 | 608
Participants | 51 | 52 | 52 | 45 | 0

14. Secondary Outcome: Percentage of Household Contacts of the Infants Born to Pregnant Women Vaccinated in Spain
Description: This analysis assessed the vaccination status of the household contacts (who accepted, received or refused vaccination) and also the reasons for refusal (not coming to site, refused to be vaccinated, unspecified) as part of an assessment of cocooning among the eligible household contacts.
Time Frame: From Day 0 (Visit 1) to Month 2 (Visit 4, end of the study).
Population: This analysis was done on the Total cohort for household contacts in Spain, which included all eligible household contacts of the infants born to pregnant women vaccinated in Spain.
Measure: Number (95% Confidence Interval); unit: Percentage of household contacts
Arm/Group | Household Group
Number analyzed (Participants) | 723
Percentage of household contacts
  Accepted vaccination | 84.4 [81.5 to 86.9]
  Received vaccination | 84.1 [81.2 to 86.7]
  Refused vaccination | 15.6 [13.1 to 18.5]
  Not coming to site | 1.4 [0.7 to 2.5]
  Refused to be vaccinated | 13.4 [11 to 16.1]
  Unspecified | 0.8 [0.3 to 1.8]

15. Secondary Outcome: Percentage of Household Contacts With SAEs
Description: SAEs assessed include medical occurrences that results in death, are life threatening, require hospitalization or prolongation of hospitalization, results in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subjects.
Time Frame: During the 31-day (Days 0-30) follow-up period post-vaccination (Boostrix administered preferably 2 weeks before the birth of the infant, Visit 3).
Population: This analysis was done on the Total cohort for household contacts which included all eligible household contacts of the infants born to pregnant women vaccinated in Spain. For the analysis of safety, all vaccinated household contacts are considered.
Measure: Number; unit: Percentage of subjects
Arm/Group | Household Group
Number analyzed (Participants) | 723
Percentage of subjects | 0

ADVERSE EVENTS:
Time Frame: For the Mothers' Groups: Solicited local and general AEs were reported during Days 0 - 7 following each dose. Unsolicited AEs were reported during Days 0 - 30 following each dose. SAEs were reported during the entire study period (Day 0 up to Month 2). For the Infants' Groups: unsolicited AEs and SAEs were reported From Day 0 (Visit 1) to Month 2 (Visit 4, end of the study). For the Household Group: SAEs were reported during the 31-day (Days 0-30) follow-up period post-vaccination.
Description: No solicited symptoms were assessed for the Infants' Groups and Household Group.
Groups:
- dTpa Group-Mother: This group consisted of pregnant women who received a single dose of Boostrix at 27-36 weeks (i.e. completed 27 weeks until 36 weeks) of gestation (Visit 1) and received a dose of the placebo post-delivery (within 72 hours).
- Control Group-Mother: This group consisted of pregnant women who received a single dose of placebo at 27-36 weeks (i.e. completed 27 weeks until 36 weeks) of gestation (Visit 1) and received a dose of Boostrix post-delivery (within 72 hours).
- Control Group-Infant: This group consisted of infants born to mothers (from Control Group Mother) who received a dose of placebo during pregnancy
Arm/Group | dTpa Group-Mother | Control Group-Mother | dTpa Group - Infant | Control Group-Infant | Household Group
All-Cause Mortality (participants affected / at risk) | 0/341 | 0/346 | 0/341 | 0/346 | 0/608
Serious Adverse Events (participants affected / at risk) | 51/341 | 52/346 | 52/341 | 45/346 | 0/608
Other Adverse Events (participants affected / at risk) | 321/341 | 303/346 | 33/341 | 29/346 | 0/608
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | dTpa Group-Mother (N=341) | Control Group-Mother (N=346) | dTpa Group - Infant (N=341) | Control Group-Infant (N=346) | Household Group (N=608)
Anaemia neonatal (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Isoimmune haemolytic disease (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial septal defect (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac septal defect (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Congenital cardiovascular anomaly (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Congenital hydronephrosis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cryptorchism (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Hypospadias (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Microtia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Polydactyly (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pyloric stenosis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syndactyly (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Transposition of the great vessels (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Trisomy 21 (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ventricular septal defect (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Hyperbilirubinaemia neonatal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 8 (8) | 6 (6) | 0 (0)
Amniotic cavity infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Beta haemolytic streptococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0)
Endometritis decidual (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mastitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neonatal infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Perineal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Sepsis neonatal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Superinfection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tracheitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac murmur (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Hypoglycaemia neonatal (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neonatal hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotonia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Somnolence neonatal (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cephalhaematoma (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Foetal distress syndrome (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Foetal growth restriction (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Hellp syndrome (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Large for dates baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Placenta praevia haemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Polyhydramnios (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 5 (5) | 7 (7) | 0 (0) | 0 (0) | 0 (0)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 11 (11) | 9 (9) | 0 (0)
Premature delivery (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Premature labour (Pregnancy, puerperium and perinatal conditions) | 11 (12) | 11 (11) | 0 (0) | 0 (0) | 0 (0)
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 13 (13) | 17 (17) | 0 (0) | 0 (0) | 0 (0)
Preterm premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Retained placenta or membranes (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small for dates baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 0 (0)
Threatened labour (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine contractions during pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vesicoureteric reflux (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Female genital tract fistula (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine atony (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Meconium aspiration syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neonatal asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neonatal respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 5 (5) | 4 (4) | 0 (0)
Transient tachypnoea of the newborn (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash neonatal (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | dTpa Group-Mother (N=341) | Control Group-Mother (N=346) | dTpa Group - Infant (N=341) | Control Group-Infant (N=346) | Household Group (N=608)
Abdominal discomfort (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 4 (5) | 1 (1) | 9 (9) | 6 (6) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Affect lability (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Afterbirth pain (Pregnancy, puerperium and perinatal conditions) | 17 (17) | 20 (20) | 0 (0) | 0 (0) | 0 (0)
Alopecia areata (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Amniotic cavity infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 11 (11) | 14 (14) | 0 (0) | 0 (0) | 0 (0)
Anaemia of pregnancy (Blood and lymphatic system disorders) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphonia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Axillary pain (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (11) | 13 (14) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast engorgement (Reproductive system and breast disorders) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Breast inflammation (Reproductive system and breast disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Cephalhaematoma (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cervical dilatation (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cervical discharge (Reproductive system and breast disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholestasis of pregnancy (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 3 (3) | 7 (8) | 3 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 8 (8) | 10 (10) | 1 (1) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 7 (7) | 0 (0) | 0 (0) | 0 (0)
Cow's milk intolerance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dacryostenosis acquired (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 4 (4) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dislocation of vertebra (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 7 (8) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eczema eyelids (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endometritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Extrapyramidal disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 188 (276) | 186 (277) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foreign body (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 6 (6) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 78 (92) | 83 (95) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 7 (7) | 6 (6) | 1 (1) | 0 (0) | 0 (0)
Genital herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Genital infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Genital infection fungal (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Granuloma (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Groin abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Grunting (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 4 (4) | 7 (7) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 129 (169) | 126 (169) | 0 (0) | 0 (0) | 0 (0)
Heart rate decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypothermia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Impaired healing (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Incision site pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site bruising (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 106 (130) | 117 (142) | 0 (0) | 0 (0) | 0 (0)
Injection site haematoma (General disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Injection site induration (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site mass (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 290 (330) | 223 (258) | 0 (0) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site rash (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 91 (101) | 92 (99) | 0 (0) | 0 (0) | 0 (0)
Injection site urticaria (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2) | 5 (5) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Labour pain (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ligament pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Mastitis (Infections and infestations) | 10 (10) | 14 (14) | 0 (0) | 0 (0) | 0 (0)
Mastitis postpartum (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Migraine with aura (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Milk allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 7 (7) | 12 (12) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nipple disorder (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nipple infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nipple inflammation (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nipple pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nodule (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 13 (13) | 0 (0) | 0 (0) | 0 (0)
Otitis media acute (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Ovarian cyst torsion (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Perineal pain (Reproductive system and breast disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Periodontitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural inflammation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural headache (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus genital (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelocaliectasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 20 (20) | 32 (33) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Raynaud's phenomenon (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Small for dates baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suppressed lactation (Reproductive system and breast disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suture related complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suture rupture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroid dysfunction in pregnancy (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinea pedis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient tachypnoea of the newborn (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Traumatic delivery (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 11 (12) | 13 (13) | 3 (3) | 1 (1) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urethral prolapse (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 8 (8) | 10 (11) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine contractions during pregnancy (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine hypotonus (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Uterine irritability (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaccination site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Varicose veins vulval (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site bruise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2015-07-15): https://cdn.clinicaltrials.gov/large-docs/49/NCT02377349/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-20): https://cdn.clinicaltrials.gov/large-docs/49/NCT02377349/SAP_001.pdf